CLINICAL TRIAL: NCT03846622
Title: Comparison of Preoperative Scoring Systems for Prediction of Perioperative Bleeding in Patients To Be Operated for Open Cardiac Surgery
Brief Title: Comparison of Scoring Systems for Bleeding in Open Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ipek Yakin Duzyol, Principal Investigator, Kocaeli Derince Education and Research Hospital
Other Study IDs: 18/34
Record Dates: First submitted 2019-01-13; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Calculation of scoring systems for bleeding

SUMMARY:
Seven different scoring systems used for prediction of perioperative bleeding were compared regarding patients operated for elective open cardiac surgery in the investigator's study.

DETAILED DESCRIPTION:
Collected data of 500 consecutive patients, operated for elective open cardiac surgery were analyzed retrospectively. Seven different scoring systems were used to predict the probability of bleeding, including TRACK, PAPWORTH, WILL-BLEED, CRUSADE, ACTION, TRUST and ACTA-PORT. The scores are calculated for each of these systems by using their own parameters, and classified into four risk groups as very low, low, moderate and high. Then, these risk groups were compared with patients identified in two groups regarding the use of perioeprative erythrocyte suspension (ES) transfusions or not, as ES positive and ES negative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 18 years of age or older,
2. Patients operated for elective open cardiac surgery.

Exclusion Criteria:

1. Patients with incomplete data,
2. Patients with an age less than 18 years,
3. Patients operated for emergent surgical procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who were operated for elective open cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Bleeding scores | Bleeding risk scores were calculated through study completion, an average of 2 years.
  Bleeding scores were calculated in points ranging from 0 to 4.(0 the lowest and 4 the highest risk score for bleeding)
The amount of blood transfusions | The amount of blood transfusions were recorded through study completion, an average of 2 years.
  The amount of blood transfusions were recorded in units.

CONTACTS AND LOCATIONS:
Overall Officials: Tolga Saracoglu, Study Director — Associate professor of the department of anaesthesiology and reanimation

IPD SHARING:
Plan to Share IPD: No